CLINICAL TRIAL: NCT05641233
Title: Preoperative Radiotherapy in Patients at High Risk of Postoperative Pancreatic Fistula After Pancreatoduodenectomy: a Multicenter Phase II Study
Brief Title: Preoperative Radiotherapy in Patients at High Risk of Postoperative Pancreatic Fistula After Pancreatoduodenectomy
Acronym: FIBROPANC-1
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Casper H.J. van Eijck, prof. dr. Casper H.J. van Eijck, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NL72913.018.20
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Neuroendocrine Carcinoma of Pancreas; Duodenum Carcinoma; Pancreas Neoplasm; Distal Cholangiocarcinoma; GIST; Pancreas Fibrosis; Pancreatic Fistula
Keywords: Post operative pancreatic fistula; Stereotactic radiotherapy; Pancreatic fibrosis; Pancreatoduodenectomy
MeSH Terms: conditions — Duodenal Neoplasms; Pancreatic Neoplasms; Pancreatic Fistula | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention arm (Experimental)
  Interventions: Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Preoperative radiotherapy delivered in a single fraction of 12 Gy focussed on 4cm pancreas at the intended (i.e. future) anastomotic site.

SUMMARY:
The FIBROPANC-1 investigates the feasibility and safety of preoperative stereotactic radiotherapy of 4cm pancreas in patients undergoing pancreatoduodenectomy at high risk (>25%) of developing post operative pancreatic fistula (POPF). A single course of 12Gy preoperative radiotherapy may lead to sufficient fibrosis in a small (4cm) targeted area, thereby reducing the risk of grade B and C POPF.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo pancreatoduodenectomy for another indication than pancreatic ductal adenocarcinoma.
* Pancreatic duct diameter ≤ 3 millimetres, measured on the diagnostic CT scan (at the level of the portomesenteric vein, at the pancreatic neck, the future anastomotic site).
* WHO-ECOG performance status 0,1 or 2.
* Ability to undergo stereotactic radiotherapy and surgery.
* Age ≥ 18 years.
* Good understanding of the oral and written patient information provided.
* Written informed consent.

Exclusion Criteria:

* Patients undergoing pancreatoduodenectomy for (suspected) pancreatic cancer, chronic pancreatitis, or benign neoplasms (e.g. serous cyst) in the periampullary region.
* Patients with (a history of) chronic pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety - CTCAE grade 3-4-5 complications related to the intervention | Up to 30 days after surgery
Hardness of pancreas texture, determined by Durometer measurement | Histopathological assesment of tissue after surgery
  Durometric measurement of the radiated and irradiated pancreatic tissue in Shore OO

SECONDARY OUTCOMES:
Percentage of patients with biochemical leak, postoperative pancreatic fistula grade B or C | Up to 30 days after operation
  Defined by the ISGPS guideline (2016)
Hardness of pancreas texture, determined intraoperatively by the pancreatic surgeon | Assesment during surgery
  Texture is scaled as soft/intermediate/hard
Macroscopic tissue assessment, determined by the pathologist | Histopathological assesment after surgery
  Evalatuation of macropscopic differences between radiated and irradiated pancreatic tissue
Surgery related postoperative complications defined according to the Clavien-Dindo classification | Up to 30 days after surgery
Overall complications | Up to 30 days after surgery
Readmission rate | Postoperative period
Length of hospital stay | Up to 30 days after surgery
  Days
30-day mortality and in-hospital mortality | Up to 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suurmeijer JA, Wismans LV, Hendriks TE, Bruynzeel AM, Nuyttens JJ, Intven MPW, van Driel LMJW, Groot Koerkamp B, Busch OR, Stoker JJ, Verheij J, Farina A, Doukas M, de Hingh IHJ, Lips DJ, van der Harst E, van Tienhoven G, Besselink MG, van Eijck CHJ; Dutch Pancreatic Cancer Group. Feasibility, safety and preliminary efficacy of preoperative stereotactic radiotherapy on the future pancreatic neck transection margin to reduce the risk of pancreatic fistula after high-risk pancreatoduodenectomy (FIBROPANC): protocol for a multicentre, single-arm trial. BMJ Open. 2024 Sep 24;14(9):e087193. doi: 10.1136/bmjopen-2024-087193. PMID 39317507